CLINICAL TRIAL: NCT06796764
Title: COMBO Endoscopy Oropharyngeal Airway Reduces Hypoxia During Sedated Gastrointestinal Endoscopy in Obese Patients: A Multicenter, Randomized, Controlled Clinical Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Diansan Su, Chair of the Department of Anesthesiology, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ZJU2025B0065
Record Dates: First submitted 2025-01-22; First posted 2025-01-28 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-08

CONDITIONS: Hypoxia; Esophageal Cancer; Gastric Cancer
Keywords: Obese Patients; The COMBO Endoscopy Oropharyngeal Airway; Hypoxia; Sedation; Gastrointestinal Endoscopy
MeSH Terms: conditions — Hypoxia; Esophageal Neoplasms; Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- the COMBO Endoscopy Oropharyngeal Airway Group (Experimental): In this group, patients use the COMBO Endoscopy Oropharyngeal Airway for oxygenation.
  Interventions: Device: the COMBO Endoscopy Oropharyngeal Airway Group
- Regular Nasal Cannula Group (Active Comparator): In this group, patients use the regular nasal cannula for oxygenation.
  Interventions: Device: Regular Nasal Cannula

INTERVENTIONS:
Device: the COMBO Endoscopy Oropharyngeal Airway Group — Using the COMBO Endoscopy Oropharyngeal Airway for oxygenation.
  Arms: the COMBO Endoscopy Oropharyngeal Airway Group
Device: Regular Nasal Cannula — Using regular nasal cannula for oxygenation.
  Arms: Regular Nasal Cannula Group

SUMMARY:
Hypoxia represents the prevailing adverse occurrence during the sedation of patients undergoing gastrointestinal endoscopy with propofol. This is particularly true for obese patients, who have a higher incidence of hypoxia. A recent innovation in this domain is the COMBO Endoscopy Oropharyngeal Airway-a multifaceted device that encompasses capnography monitoring, bite block , oxygenation support, and oropharyngeal airway management. This device has been purposefully designed to cater to the unique requirements of endoscopic procedures. The principal objective of this study is to assess the efficacy and safety of the COMBO Endoscopy Oropharyngeal Airway in reducing the incidence of hypoxia in obese patients undergoing gastrointestinal endoscopy under sedation.

ELIGIBILITY:
Inclusion Criteria:

* Age 18≤ Age ≤70.
* BMI ≥ 28 kg/m².
* The ASA classification ranges from I to II.
* Patients have signed the informed consent form.
* Patients undergoing gastroendoscopy and colonoscopy procedure.
* The estimated duration of the procedure does not exceed 45 minutes.

Exclusion Criteria:

* Patients who exhibit contraindications to oropharyngeal airway ventilation, such as coagulation disorders, a predisposition to oral and nasal bleeding, mucosal damage, or anatomical constraints impeding oropharyngeal channel placement.
* Severe cardiac insufficiency, defined as a maximal exercise capacity of less than 4 metabolic equivalents (METs).
* Profound renal insufficiency necessitating preoperative dialysis.
* A confirmed severe liver dysfunction.
* Patients diagnosed with chronic obstructive pulmonary disease (COPD) or those presently experiencing other acute and chronic pulmonary conditions necessitating prolonged or intermittent oxygen therapy.
* Elevated intracranial pressure.
* Upper respiratory tract infections, encompassing the oral, nasal, and pharyngeal regions.
* Fever, defined as a core body temperature exceeding 37.5 degrees Celsius.
* Pregnancy or lactation.
* Hypersensitivity reactions to sedatives like propofol or medical equipment such as adhesive tape.
* Urgent surgical intervention.
* Polytrauma.
* Peripheral oxygen saturation (SpO2) levels below 95% while breathing room air preoperatively.
* BMI<28 kg/m².
* Patients with a documented history of substance abuse, specifically drugs and/or alcohol, within the two years preceding the commencement of the screening period. Substance abuse in this context is defined as consuming more than three standard alcoholic beverages daily, roughly equivalent to 10g of alcohol or 50g of Chinese Baijiu.
* Patients with a history of mental and neurological disorders, including but not limited to depression, severe central nervous system depression, Parkinson's disease, basal ganglia lesions, schizophrenia, epilepsy, Alzheimer's disease, and myasthenia gravis.
* Presently engaged in concurrent participation in additional clinical trials.
* Patients considered ineligible by researchers for inclusion in this clinical trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 580 (Estimated)
Dates: Start 2025-04-11 (Actual); Primary Completion 2025-12-04 (Estimated); Study Completion 2025-12-04 (Estimated)

PRIMARY OUTCOMES:
The incidence of hypoxia | Patients will be followed for the duration of hospital stay, an expected average about 2 hours
  75% ≤ SpO2 < 90% for <60 s

SECONDARY OUTCOMES:
The incidence of sub-clinical respiratory depression | Patients will be followed for the duration of hospital stay, an expected average about 2 hours
  90% ≤ SpO2 < 95%
SpO2 < 75% or 75% ≤ SpO2 < 90% for ≥60 s | Patients will be followed for the duration of hospital stay, an expected average about 2 hours
  SpO2 < 75% or 75% ≤ SpO2 < 90% for ≥60 s

OTHER OUTCOMES:
The incidence of other adverse events | Patients will be followed for the duration of hospital stay, an expected average about 2 hours
  Other adverse events recorded by tools proposed by the World Society of Intravenous Anesthesia International Sedation Task Force

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The Fourth Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Cancer hospital, Hangzhou, Zhejiang